CLINICAL TRIAL: NCT04429997
Title: Prospective Randomized Controlled Trial: Comparison of Incidence of Patellar Crepitus Between Removal and Non-removal of Fibrosynovial Tissue at the Border of the Superior Pole of the Patellar
Brief Title: Incidence of Patellar Crepitus in Removal and Non-removal of Fibrosynovial Tissue at Superior Pole of Patella
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: COA 057/2563
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Removal of Fibrosynovial Tissue; Non-removal of Fibrosynovial Tissue; Patellar Non-resurfacing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removal of fibrosynovial tissue (Experimental): Removal of fibrosynovial tissue in patellar non-resurfacing TKA
  Interventions: Procedure: Removal of fibrosynovial tissue
- Non-removal of fibrosynovial tissue (Experimental): Non-removal of fibrosynovial tissue in patellar non-resurfacing TKA
  Interventions: Procedure: Non-removal of fibrosynovial tissue

INTERVENTIONS:
Procedure: Removal of fibrosynovial tissue — Remove of fibrosynovial tissue at the superior border of patella
  Arms: Removal of fibrosynovial tissue
Procedure: Non-removal of fibrosynovial tissue — Do not remove of fibrosynovial tissue at the superior border of patella
  Arms: Non-removal of fibrosynovial tissue

SUMMARY:
The purpose of this study is to compare the incidence of patellar crepitus complication and the clinical outcome between remove and not remove fibrosynovial tissue at the border of the superior pole of the patellar in posterior stabilized total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee who were scheduled for a primary total knee arthroplasty

Exclusion Criteria:

* Valgus deformity
* History of inflammatory arthroplathy
* Previous fracture or open surgery on the same knee
* History of patellar instability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of patellar crepitus complication | Change from baseline patellar crepitus complication 3 months, 6 months, and 12 months after surgery
  Incidence of patellar crepitus complication (present, absent)

SECONDARY OUTCOMES:
Knee Society and Knee Society function score | Change from baseline Knee Society and Knee Society function score at 3 months, 6 months, and 12 months after surgery
  Knee Society and Knee Society function score (minimum 0, maximum 200)
New patellar score | Change from baseline new patellar score at 3 months, 6 months, and 12 months after surgery
  New patellar score (minimum 0, maximum 30)
Oxford knee score | Change from baseline Oxford knee score 3 months, 6 months, and 12 months after surgery
  Oxford knee score (minimum 0, maximum 48)
Change of post-operative anterior knee pain | Change from baseline Visual Analog Scale for anterior knee pain at 3 months, 6 months, and 12 months after surgery
  Visual Analog Scale for anterior knee pain (minimum 0, maximum 10) Do higher values represent a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Department of Orthopaedics, Faculty of Medicine Vajira Hospital, Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand